CLINICAL TRIAL: NCT02343094
Title: Phenylbutyrate Effect on Lcn2 Urianry Expression in Proteinuric Patients
Brief Title: Phenylbutyrate in Proteinuric Nephropathies
Acronym: PIRATE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-003924-35
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Proteinuric Diseases
Keywords: Proteinuria; Lipocalin 2; Neutrophil gelatinase associated lipocalin; ELISA
MeSH Terms: conditions — Proteinuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PBA 7,5g/d (Experimental): Treatment for 14 days
  Interventions: Drug: PBA 7,5g/d
- PBA 15g/d (Experimental): Treatment for 14 days
  Interventions: Drug: PBA 15g/d

INTERVENTIONS:
Drug: PBA 7,5g/d — Treatment for 14 days with PBA
  Arms: PBA 7,5g/d
Drug: PBA 15g/d — Treatment for 14 days with PBA
  Arms: PBA 15g/d

SUMMARY:
The purpose of this study is to determine whether sodium phenylbutyrate can reduce Lcn2 urinary expression in proteinuric patients.

DETAILED DESCRIPTION:
Proteinuria is a major prognosis factor of chronic kidney disease (CKD) progression. Convergent evidences from clinical and experimental studies indicate that albuminuria and proteinuria are not simply a marker of CKD progression, but an active player in the evolution of the disease. Mechanistically, it has been shown that proteinuria induces endoplasmic reticulum stress in tubular cells, leading to induction of lipocalin 2/NGAL, a critical element of CKD progression. Moreover, proteinuric mice treated with phenylbutyrate are protected from CKD progression.

The aim of this study is to evaluate the efficacy of phenybutyrate, a molecular chaperone which inhibits ER stress, on the proteinuria-induced NGAL expression. Urinary NGAL/creatinine ratio will be evaluated in proteinuric patients before and under treatment with phenylbutyrate.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney disease for ore than 3 months
* Proteinuria > 1g/d or 0,1g/mmmol creatinine
* eGFR >30ml/mn/1,73m2
* written informed consent
* affiliated with social security health insurance

Exclusion Criteria:

* Women with childbearing potential
* Recent (<3 months) modification of ACE inhibitors or ARB
* Acute renal failure
* eGFR <30ml/mn/1,73m2
* Nephrotic syndrome (albuminélia <30g/l)
* Infection with HIV, HCV, HBV
* Liver insufficiency
* No affiliated with social security health insurance
* inclusion in another protocol of biomedical research
* risk of non-adherence to protocol and visits
* patients having a cardiac insufficiency of grade 3 or 4
* patient requiring of a strict salt-free diet
* patients under corticoids or immunosuppresseurs
* clinical intolerance in the treatment
* intolerance in the fructose, the syndrome of malabsorption glucose and galactose or a deficit in sucrase / isomaltase
* patients treated by Probenecide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Urinary Lcn2/creatinine ratio | Day 7, Day 15, Day 21, Day 28
  Reduction of 50 % of Lcn2 concentration, measured with ELISA

SECONDARY OUTCOMES:
Urinary protein/creatinine ratio | Day 7
  Reduction of 30% of the proteinurie and the albuminuria
Urinary protein/creatinine ratio | Day 15
  Reduction of 30% of the proteinurie and the albuminuria
Urinary protein/creatinine ratio | Day 21
  Reduction of 30% of the proteinurie and the albuminuria
Urinary protein/creatinine ratio | Day 28
  Reduction of 30% of the proteinurie and the albuminuria

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand KNEBELMANN, Principal Investigator — Service de Néphrologie Adulte, Hôpital Necker
Locations (1):
- Hôpital Necker Enfants Malades, Paris, France